CLINICAL TRIAL: NCT03326128
Title: High Dose Bupropion Treatment for Smoking Cessation - Pilot Study
Brief Title: High Dose Bupropion for Smoking Cessation - Pilot Study
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to the COVID-19 pandemic, it was difficult to recruit eligible participants.
Sponsor: University of Southern California (Other)
Collaborators: University of California, Los Angeles (Other); University of California, San Diego (Other)
Responsible Party: Principal Investigator, Adam Leventhal, Associate Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1703346
Record Dates: First submitted 2017-10-18; First posted 2017-10-31 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Smoking Cessation; Smoking, Tobacco; Smoking (Tobacco) Addiction; Cessation, Tobacco; Cigarette Smoking
Keywords: Bupropion; Smokers; Smoking cessation; Cigarette smoking; Cigarette
MeSH Terms: conditions — Smoking Cessation; Tobacco Smoking; Smoking; Behavior, Addictive; Tobacco Use Cessation; Cigarette Smoking | interventions — Bupropion

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to receive either 300 or 450 mg of Bupropion.
Who Masked: Participant
Masking Description: Participants will be unaware of which medication condition they have been assigned to; however, the study team and the care provider will know which dose of medication they are distributing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BUP-300 (Active Comparator): Participants will receive Bupropion hydrochloride for 10 weeks and titrate to a maximum dose of 300 mg/day and will also receive standard smoking cessation counseling for 8 weeks.
  Interventions: Drug: Bupropion Hydrochloride
- BUP-450 (Experimental): Participants will receive Bupropion hydrochloride for 12 weeks and titrate to a maximum dose of 450 mg/day and will also receive standard smoking cessation counseling for 8 weeks.
  Interventions: Drug: Bupropion Hydrochloride

INTERVENTIONS:
Drug: Bupropion Hydrochloride — Antidepressant that is also effective in smoking cessation
  Other Names: Bupropion

SUMMARY:
This study aims to investigate the benefit of administering two differing doses of Bupropion (BUP) to smokers to assist with smoking cessation.

DETAILED DESCRIPTION:
Participants will be randomly assigned to either receive 300 mg of BUP or 450 mg of BUP for 8 weeks with an aim to quit smoking. In addition, participants will simultaneously receive counseling to set a quit date and stay motivated to quit. Medication will be administered up to 4 weeks before and for 4 weeks after designated quit-date. Post-treatment follow-up appointment will be scheduled for 8, 16, and 26 weeks post treatment to assess commitment to quitting and overall success of the study.

ELIGIBILITY:
Inclusion Criteria:

* Smokes cigarettes daily for at least 1 year
* Breath CO of 5 ppm or higher at Baseline visit
* Age 21 - 65

Exclusion Criteria:

* Possible drug contraindications (panic disorder, bipolar disorder, bulimia, anorexia, insomnia, suicidal ideation, alcohol withdrawal, seizures, severe hypertension, renal/hepatic impairment, angle closure glaucoma)
* Unstable cardiovascular disorder or uncontrolled hypertension
* Severe renal/hepatic impairment based on serology evaluation
* History of seizures, liver failure, central nervous system tumor, central nervous system infection, hypoglycemia, hyponatremia, hypoxia, stroke arteriovenous malformation, head injury
* Current use of other cessation medication or counseling
* History of bupropion use
* Current anti-psychotic, anxiolytic, antidepressant, or psychostimulant medication use, other drugs that may lower seizure threshold, CYP2B6 inhibitors, CYP2B6 inducers, drug metabolized by CYP2D6
* Sudden stoppage of alcohol, benzodiazepines, barbiturates, or antiepileptic drugs
* Current (past 30 days) use of illicit or medical use of prescription stimulants
* Currently or plan to be pregnant or breastfeeding

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Point Prevalence Abstinence (PPA) [change in abstinence reports will be assessed] | Through study completion, an average of 26 months
  Self report of smoking status

SECONDARY OUTCOMES:
Smoking cessation milestones | Through study completion, an average of 26 months
  Smoking timeline follow back interview
Inventory of Depressive and Anxious Symptomology (General depression subscale) | Through study completion, an average of 26 months
  This measure is obtained through the completion of the Inventory of Depressive and Anxious Symptomology General depression subscale. A total score will be calculated. Scores can range from 4 to 20 with the lower scores representing lower levels of depression and higher scores representing higher levels of depression.
Inventory of Depressive and Anxious Symptomology (Social anxiety subscale) | Through study completion, an average of 26 months
  This measure is obtained through the completion of the Inventory of Depressive and Anxious Symptomology Social anxiety subscale. A total score will be calculated. Scores can range from 4 to 20 with the lower scores representing lower levels of social anxiety and higher scores representing higher levels of social anxiety.
Inventory of Depressive and Anxious Symptomology (Traumatic intrusions subscale) | Through study completion, an average of 26 months
  This measure is obtained through the completion of the Inventory of Depressive and Anxious Symptomology Traumatic intrusions subscale. A total score will be calculated. Scores can range from 4 to 20 with the lower scores representing fewer traumatic intrusions and g scores representing greater traumatic intrusions.
Self report scale for Attention deficit/Hyperactivity disorder (ADHD) | Baseline visit
  ADHD symptom report
Snaithe-Hamilton Pleasure Scale (SHAPS) | Baseline visit and Week 8 post quit date
  Anhedonia scale
Objective body weight | Baseline visit and Week 8 post quit date
  Measured with a medical grade scale
Body adiposity via bioimpedence monitor | Baseline visit and Week 8 post quit date
  Measures body fat percentage/ BMI

CONTACTS AND LOCATIONS:
Overall Officials: Adam M Leventhal, PhD, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leventhal AM, Kahler CW, Ray LA, Zimmerman M. Refining the depression-nicotine dependence link: patterns of depressive symptoms in psychiatric outpatients with current, past, and no history of nicotine dependence. Addict Behav. 2009 Mar;34(3):297-303. doi: 10.1016/j.addbeh.2008.11.008. Epub 2008 Nov 21. PMID 19062199
- [Background] Brown RA, Niaura R, Lloyd-Richardson EE, Strong DR, Kahler CW, Abrantes AM, Abrams D, Miller IW. Bupropion and cognitive-behavioral treatment for depression in smoking cessation. Nicotine Tob Res. 2007 Jul;9(7):721-30. doi: 10.1080/14622200701416955. PMID 17577801
- [Background] Fava M, Rush AJ, Thase ME, Clayton A, Stahl SM, Pradko JF, Johnston JA. 15 years of clinical experience with bupropion HCl: from bupropion to bupropion SR to bupropion XL. Prim Care Companion J Clin Psychiatry. 2005;7(3):106-13. doi: 10.4088/pcc.v07n0305. PMID 16027765
- [Background] Ameringer KJ, Chou CP, Leventhal AM. Shared versus specific features of psychological symptoms and cigarettes per day: structural relations and mediation by negative- and positive-reinforcement smoking. J Behav Med. 2015 Apr;38(2):224-36. doi: 10.1007/s10865-014-9597-y. Epub 2014 Sep 18. PMID 25231408
- [Background] Leventhal AM, Mickens L, Dunton GF, Sussman S, Riggs NR, Pentz MA. Tobacco use moderates the association between major depression and obesity. Health Psychol. 2010 Sep;29(5):521-8. doi: 10.1037/a0020854. PMID 20836607
- [Background] Boutelle KN, Monreal T, Strong DR, Amir N. An open trial evaluating an attention bias modification program for overweight adults who binge eat. J Behav Ther Exp Psychiatry. 2016 Sep;52:138-146. doi: 10.1016/j.jbtep.2016.04.005. Epub 2016 Apr 16. PMID 27116704
- [Background] Boutelle KN, Braden A, Douglas JM, Rhee KE, Strong D, Rock CL, Wilfley DE, Epstein L, Crow S. Design of the FRESH study: A randomized controlled trial of a parent-only and parent-child family-based treatment for childhood obesity. Contemp Clin Trials. 2015 Nov;45(Pt B):364-370. doi: 10.1016/j.cct.2015.09.007. Epub 2015 Sep 8. PMID 26358536
- [Background] Boutelle KN, Liang J, Knatz S, Matheson B, Risbrough V, Strong D, Rhee KE, Craske MG, Zucker N, Bouton ME. Design and implementation of a study evaluating extinction processes to food cues in obese children: the Intervention for Regulations of Cues Trial (iROC). Contemp Clin Trials. 2015 Jan;40:95-104. doi: 10.1016/j.cct.2014.11.011. Epub 2014 Nov 22. PMID 25461494
- [Background] Ebbert JO, Hatsukami DK, Croghan IT, Schroeder DR, Allen SS, Hays JT, Hurt RD. Combination varenicline and bupropion SR for tobacco-dependence treatment in cigarette smokers: a randomized trial. JAMA. 2014 Jan 8;311(2):155-63. doi: 10.1001/jama.2013.283185. PMID 24399554
- [Background] Leventhal AM, Munafo M, Tidey JW, Sussman S, Monterosso JR, Sun P, Kahler CW. Anhedonia predicts altered processing of happy faces in abstinent cigarette smokers. Psychopharmacology (Berl). 2012 Jul;222(2):343-51. doi: 10.1007/s00213-012-2649-5. Epub 2012 Feb 4. PMID 22311383
- [Background] Leventhal AM, Trujillo M, Ameringer KJ, Tidey JW, Sussman S, Kahler CW. Anhedonia and the relative reward value of drug and nondrug reinforcers in cigarette smokers. J Abnorm Psychol. 2014 May;123(2):375-86. doi: 10.1037/a0036384. PMID 24886011
- [Background] Leventhal AM, Ameringer KJ, Osborn E, Zvolensky MJ, Langdon KJ. Anxiety and depressive symptoms and affective patterns of tobacco withdrawal. Drug Alcohol Depend. 2013 Dec 1;133(2):324-9. doi: 10.1016/j.drugalcdep.2013.06.015. Epub 2013 Jul 26. PMID 23896304

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-25): https://cdn.clinicaltrials.gov/large-docs/28/NCT03326128/Prot_SAP_000.pdf